CLINICAL TRIAL: NCT03596840
Title: Effectiveness of Different Antihypertensive Medications on Urine Albumin-to-Creatinine Ratio (UACR) in Community Hypertensive Patients With Microalbuminuria
Brief Title: Community-based Microalbuminuria Screening in Patients With Hypertension
Acronym: CMSIH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xuejuan Jin, Associate Professor, Shanghai Zhongshan Hospital
Other Study IDs: B2018-106
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hypertension; Microalbuminuria
Keywords: Hypertension; Microalbuminuria; Effectiveness; Antihypertensive medications
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the effectiveness of different anti-hypertensive drugs on patients with hypertension and microalbuminuria.

DETAILED DESCRIPTION:
This is a a real world registry study. All patients with hypertension in community hospitals in China will be eligible . Patient demographics, medical history, clinical characteristics, physical examination, laboratory tests (including UCAR, blood routine, urine routine, blood biochemistry, and ECG), antihypertensive drugs (including: ACEI/ ARB, thiazide diuretics, CCB, beta-blockers, alpha-blockers, and other antihypertensive drugs used in real-life clinical practice in other communities.) will be recorded. All patients are anticipated to be followed up for 12-month. Effectiveness of different antihypertensive medications on Urine Albumin-to-Creatinine Ratio (UACR) will be evaluted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension;
* Urinary albumin/creatinine ratio in random urine samples is 30-300 mg/g
* Age >=18
* Understand and sign informed consent

Exclusion Criteria:

* This is a real-world registry study and does not set exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Hypertensive Patients With Microalbuminuria
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Urine Albumin-to-Creatinine Ratio (UCAR) | 12 months
  Differences in UCAR between with ACEI/ARB and without ACEI/ARB

SECONDARY OUTCOMES:
Combined endpoints: re-admission, cardiovascular events, and all-cause mortality | 12 months
  Differences in Combined endpoints between with ACEI/ARB and without ACEI/ARB